CLINICAL TRIAL: NCT01325428
Title: An Open Label, Phase II Trial of Afatinib With or Without Vinorelbine for the Treatment of HER2-overexpressing Inflammatory Breast Cancer
Brief Title: Afatinib (BIBW2992) in HER2 (Human Epidermal Growth Factor Receptor 2)-Overexpressing Inflammatory Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.89; 2010-024454-10 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- Afatinib once daily (OD) (Experimental): Patients receive afatinib monotherapy once daily until progression of their disease
  Interventions: Drug: Afatinib once daily (OD); Drug: Vinorelbine Weekly

INTERVENTIONS:
Drug: Afatinib once daily (OD) — Patient to receive afatinib monotherapy until progression of their disease
Drug: Vinorelbine Weekly — Patients additionally receive vinorelbine weekly on disease progression on afatinib monotherapy

SUMMARY:
The general aim of this study is to investigate the efficacy and safety of afatinib alone and in combination with weekly vinorelbine (in patients who progress on afatinib monotherapy within this trial) as treatment in patients with HER2-overexpressing, locally advanced or metastatic inflammatory breast cancer. The study will include patients who have and have not failed prior trastuzumab treatment.

ELIGIBILITY:
Inclusion criteria:

1. Female patients >=18 years with proven diagnosis of HER2-overexpressing, histologically confirmed breast cancer
2. Locally advanced or metastatic disease
3. Must have disease that can be evaluated according to RECIST 1.1 (Response Evaluation Criteria for Solid Tumours version 1.1)
4. For trastuzumab pre-treated patients, must have failed prior trastuzumab treatment
5. Investigator-confirmed diagnosis of Inflammatory Breast Cancer
6. Must have biopsiable disease

Exclusion criteria:

1. Prior treatment with HER2-targeted small molecules or antibodies other than trastuzumab (which must have been given in the trastuzumab-failure study population)
2. Must not have received prior vinorelbine treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (16):
- United States (2):
  - 1200.89.10001 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1200.89.10005 Boehringer Ingelheim Investigational Site, Durham, North Carolina
- Australia (2):
  - 1200.89.61002 Boehringer Ingelheim Investigational Site, East Bentleigh, Victoria
  - 1200.89.61003 Boehringer Ingelheim Investigational Site, Perth, Western Australia
- 1200.89.85201 Boehringer Ingelheim Investigational Site, Hong Kong, Hong Kong
- South Korea (2):
  - 1200.89.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1200.89.82002 Boehringer Ingelheim Investigational Site, Seoul
- Thailand (4):
  - 1200.89.66002 Boehringer Ingelheim Investigational Site, Bangkok
  - 1200.89.66004 Boehringer Ingelheim Investigational Site, Bangkok
  - 1200.89.66003 Boehringer Ingelheim Investigational Site, Chiang Mai
  - 1200.89.66001 Boehringer Ingelheim Investigational Site, Hat-Yai, Songkhla
- Tunisia (2):
  - 1200.89.21601 Boehringer Ingelheim Investigational Site, Aryanah
  - 1200.89.21602 Boehringer Ingelheim Investigational Site, Sousse
- United Kingdom (3):
  - 1200.89.44002 Boehringer Ingelheim Investigational Site, Bournemouth
  - 1200.89.44001 Boehringer Ingelheim Investigational Site, London
  - 1200.89.44003 Boehringer Ingelheim Investigational Site, London

REFERENCES:
- [Derived] Goh G, Schmid R, Guiver K, Arpornwirat W, Chitapanarux I, Ganju V, Im SA, Kim SB, Dechaphunkul A, Maneechavakajorn J, Spector N, Yau T, Afrit M, Ahmed SB, Johnston SR, Gibson N, Uttenreuther-Fischer M, Herrero J, Swanton C. Clonal Evolutionary Analysis during HER2 Blockade in HER2-Positive Inflammatory Breast Cancer: A Phase II Open-Label Clinical Trial of Afatinib +/- Vinorelbine. PLoS Med. 2016 Dec 6;13(12):e1002136. doi: 10.1371/journal.pmed.1002136. eCollection 2016 Dec. PMID 27923043

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study conducted in two sequential parts (Part A in which patients were treated with Afatinib (BIBW 2992) as monotherapy; Part B in which patients were treated with Afatinib plus Vinorelbine as combination therapy after progression on Afatinib monotherapy).
Pre-assignment Details: Part A: Patients were treated with Afatinib and could continue on treatment until first Progression of Disease (PD), intolerable side effects, or withdrawal of consent. Upon first PD, patients could enter Part B of the study, during which they continued to be treated with Afatinib and additionally were treated with weekly Vinorelbine.
Groups:
- Afatinib (Part A). Afatinib+V (Vinorelbine) (Part B).: Part A: Patients received Afatinib tablets, 40 mg taken orally Once Daily (OD) until Progression of their Disease (PD). In case of treatment-related adverse events (AEs), the 40 mg dose could be reduced by increments of 10 mg to 30 mg once daily or 20 mg once daily.
  Part B: Upon first Progression of Disease (PD), patients could enter Part B of the study, during which they continued to be treated with Afatinib and additionally were treated with Vinorelbine 25 mg/m2 per week via intravenous (i.v) infusion. Patients treated with Afatinib and Vinorelbine combination therapy could continue to receive treatment until second progression of disease, intolerable side effects, or withdrawal of consent.
Period: Part A
Arm/Group | Afatinib (Part A). Afatinib+V (Vinorelbine) (Part B).
Started | 26
Completed | 10
Not Completed | 16
Not completed — Progressive disease according to RECIST | 9
Not completed — Clinical signs, symptoms of progression | 2
Not completed — Other adverse event | 1
Not completed — Refused continue taking trial medication | 2
Not completed — Other reason not defined above | 2
Period: Part B
Arm/Group | Afatinib (Part A). Afatinib+V (Vinorelbine) (Part B).
Started | 10
Completed | 7
Not Completed | 3
Not completed — Refused continue taking trial medication | 2
Not completed — Other reason not defined above | 1

BASELINE CHARACTERISTICS:
Population: TRT A Treated set (Part A): All patients who were documented to have taken at least one dose of Afatinib in Part A.
  TRT B Treated set (Part B): All patients who received at least one dose each of Afatinib and Vinorelbine in Part B.
Groups:
- Part A: Afatinib Once Daily. Part B: Afatinib+V (Vinorelbine).: Part A: Patients received Afatinib tablets, 40 mg taken orally Once Daily (OD) until Progression of their Disease (PD). In case of treatment-related AEs, the 40 mg dose could be reduced by increments of 10 mg to 30 mg once daily or 20 mg once daily.
  Part B: Upon first Progression of Disease (PD), patients could enter Part B of the study, during which they continued to be treated with Afatinib and additionally were treated with Vinorelbine 25 mg/m2 per week via intravenous (i.v) infusion. Patients treated with Afatinib and Vinorelbine combination therapy could continue to receive treatment until second progression of disease, intolerable side effects, or withdrawal of consent.
Arm/Group | Part A: Afatinib Once Daily. Part B: Afatinib+V (Vinorelbine).
Number analyzed (Participants) | 26
Age, Customized [Mean (Standard Deviation); unit: Years]
  Part A | 51.5 (8.8)
  Part B | 51.5 (12.5)
Sex/Gender, Customized [Number; unit: Participants]
  Female (Part A) | 26
  Female (Part B) | 10
  Male (Part A) | 0
  Male (Part B) | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Clinical Benefit (CB) Assessed by Complete Response (CR), Partial Response (PR) or Stable Disease (SD) for at Least 6 Months Using the Response Evaluation Criteria in Solid Tumours (RECIST 1.1).
Description: Tumour response was assessed separately for Part A and Part B according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The primary endpoint of this study was confirmed clinical benefit, as assessed by Stable Disease (SD) for at least 6 months (defined as >182 days), Partial Response (PR), or Complete Response (CR) according to RECIST version 1.1 (only confirmed responses were considered).
Time Frame: This endpoint was assessed between the from first administration of trial medication in Part A and the earliest of PD, death or start of next treatment (either Part B combination therapy or new anti-cancer therapy) up to 929 days.
Population: TRT A Treated Set (Part A): All patients who were documented to have taken at least one dose of Afatinib in Part A.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part A: Afatinib Once Daily (OD).: Part A: Patients received Afatinib tablets, 40 mg taken orally Once Daily (OD) until PD. In case of treatment-related AEs, the 40 mg dose could be reduced by increments of 10 mg to 30 mg once daily or 20 mg once daily.
  The 95% Confidence Interval is Exact Confidence Interval.
Arm/Group | Part A: Afatinib Once Daily (OD).
Number analyzed (Participants) | 26
Percentage of participants | 35 [17 to 56]

2. Primary Outcome: Part B: Clinical Benefit (CB) Assessed by Complete Response (CR), Partial Response (PR) or Stable Disease (SD) for at Least 6 Months Using the Response Evaluation Criteria in Solid Tumours (RECIST 1.1).
Description: Tumour response was assessed separately for Part B according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The primary endpoint of this study was confirmed clinical benefit, as assessed by Stable Disease (SD) for at least 6 months (defined as >182 days), Partial Response (PR), or Complete Response (CR) according to RECIST version 1.1 (only confirmed responses were considered).
Time Frame: This endpoint was recorded from first administration of trial medication in Part B until the earliest of PD, death or start of new anti-cancer therapy up to 929 days.
Population: TRT B Treated set (Part B): All patients who received at least one dose each of Afatinib and Vinorelbine in Part B.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part B: Afatinib Once Daily (OD)+V (Vinorelbine).: Part B: Upon first Progression of Disease (PD), patients could enter Part B of the study, during which they continued to be treated with Afatinib and additionally were treated with Vinorelbine 25 mg/m2 per week via intravenous (i.v) infusion. Patients treated with Afatinib and Vinorelbine combination therapy could continue to receive treatment until second progression of disease, intolerable side effects, or withdrawal of consent. The 95% Confidence Interval is Exact Confidence Interval.
Arm/Group | Part B: Afatinib Once Daily (OD)+V (Vinorelbine).
Number analyzed (Participants) | 10
Percentage of participants | 20 [3 to 56]

3. Secondary Outcome: Part A: Confirmed Objective Response (OR) Assessed by Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST 1.1).
Description: Objective response was defined on a patient level as a best response of CR or PR.
Time Frame: This endpoint was recorded from first administration of trial medication until the earliest of disease progression, death or start of next treatment (either Part B combination therapy or new anti-cancer therapy) up to 929 days.
Population: TRT A Treated Set (Part A): All patients who were documented to have taken at least one dose of Afatinib in Part A.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part A: Afatinib Once Daily (OD).: Part A: Patients received Afatinib tablets, 40 mg taken orally Once Daily (OD) until progression of their disease. In case of treatment-related AEs, the 40 mg dose could be reduced by increments of 10 mg to 30 mg once daily or 20 mg once daily. The 95% Confidence Interval is Exact Confidence Interval.
Arm/Group | Part A: Afatinib Once Daily (OD).
Number analyzed (Participants) | 26
Percentage of participants | 31 [14 to 52]

4. Secondary Outcome: Part B: Confirmed Objective Response (OR) Assessed by Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST 1.1).
Description: Objective response was defined on a patient level as a best response of CR or PR.
Time Frame: This endpoint was recorded from first administration of trial medication in Part B and until the earliest of disease progression, death or start of new anti-cancer therapy up to 929 days.
Population: TRT B Treated set (Part B): All patients who received at least one dose each of Afatinib and Vinorelbine in Part B.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Afatinib Once Daily (OD)+V (Vinorelbine).
Number analyzed (Participants) | 10
Percentage of participants | 10 [0 to 45]

5. Secondary Outcome: Part A: Unconfirmed Objective Response (OR) Assessed by Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST 1.1).
Description: Objective response was defined on a patient level as a best response of CR or PR.
Time Frame: This endpoint was recorded from first administration of trial medication until the earliest of PD, death or start of next treatment (either Part B combination therapy or new anti-cancer therapy) up to 929 days.
Population: TRT A Treated Set (Part A): All patients who were documented to have taken at least one dose of Afatinib in Part A.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: Afatinib Once Daily (OD).
Number analyzed (Participants) | 26
Percentage of participants | 42 [23 to 63]

6. Secondary Outcome: Part B: Unconfirmed Objective Response (OR) Assessed by Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST 1.1 ).
Description: Objective response was defined on a patient level as a best response of CR or PR.
Time Frame: This endpoint was recorded from first administration of trial medication in Part B and until the earliest of PD, death or start of new anti-cancer therapy up to 929 days.
Population: TRT B Treated set (Part B): All patients who received at least one dose each of Afatinib and Vinorelbine in Part B.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Afatinib Once Daily (OD)+V (Vinorelbine).
Number analyzed (Participants) | 10
Percentage of participants | 30 [7 to 65]

7. Secondary Outcome: Part A: Duration of Unconfirmed Objective Response.
Description: Objective Response (OR) was defined on a patient level as a best response of Complete Response (CR) or Partial Response (PR). Duration of objective response was measured from the time of first unconfirmed objective response to the time of progression or death (or date of censoring for Progression Free Survival (PFS)).
Time Frame: From first drug administration until end of Part A, up to 929 days.
Population: TRT A Treated Set (Part A): All patients who were documented to have taken at least one dose of Afatinib in Part A.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Part A: Afatinib Once Daily (OD).: Part A: Patients received Afatinib tablets, 40 mg taken orally Once Daily (OD) until progression of their disease. In case of treatment-related AEs, the 40 mg dose could be reduced by increments of 10 mg to 30 mg once daily or 20 mg once daily.
Arm/Group | Part A: Afatinib Once Daily (OD).
Number analyzed (Participants) | 11
Days | NA [57 to NA] — The Kaplan Meier (KM) probability never falls to 0.5 therefore the median can't be estimated. Not Applicable (NA).

8. Secondary Outcome: Part B: Duration of Unconfirmed Objective Response.
Description: Objective response was defined on a patient level as a best response of CR or PR. Duration of objective response was measured from the time of first unconfirmed objective response to the time of progression or death (or date of censoring for PFS).
Time Frame: From first drug administration until end of Part B, up to 929 days.
Population: TRT B Treated set (Part B): All patients who received at least one dose each of Afatinib and Vinorelbine in Part B.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part B: Afatinib Once Daily (OD)+V (Vinorelbine).
Number analyzed (Participants) | 3
Days | 57 [56 to 140]

9. Secondary Outcome: Part A: Progression Free Survival.
Description: PD was evaluated according to the RECIST version 1.1. For patients with a known date of progression (or death), PFS was the earlier of date of progression or death - date of first administration + 1. The date of progression and date of first administration referred to the respective part of the study A.
Time Frame: From first drug administration until end of Part A, up to 713 days.
Population: TRT A Treated Set (Part A): All patients who were documented to have taken at least one dose of Afatinib in Part A.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part A: Afatinib Once Daily (OD).
Number analyzed (Participants) | 26
Days | 110.5 [58.0 to 386.0]

10. Secondary Outcome: Part B: Progression Free Survival.
Description: PD was evaluated according to the RECIST version 1.1. For patients with a known date of progression (or death), PFS was the earlier of date of progression or death - date of first administration + 1. The date of progression and date of first administration referred to the respective part of the study B.
Time Frame: From first drug administration until end of Part B, up to 230 days.
Population: TRT B Treated set (Part B): All patients who received at least one dose each of Afatinib and Vinorelbine in Part B.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part B: Afatinib Once Daily (OD)+V (Vinorelbine).
Number analyzed (Participants) | 10
Days | 106.0 [36.0 to 190.0]

11. Secondary Outcome: Progression Free Survival Over the Whole Sudy.
Description: PD was evaluated according to the RECIST version 1.1. Number of days from the start of monotherapy to the date of second PD.
Time Frame: From first drug administration until end of study, up to 700 days.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Afatinib Once Daily (OD). Afatinib+V (Vinorelbine).: Part A: Patients received Afatinib tablets, 40 mg taken orally Once Daily (OD) until PD. In case of treatment-related AEs, the 40 mg dose could be reduced by increments of 10 mg to 30 mg once daily or 20 mg once daily.
  Part B: Upon first Progression of Disease (PD), patients could enter Part B of the study, during which they continued to be treated with Afatinib and additionally were treated with Vinorelbine 25 mg/m2 per week via intravenous (i.v) infusion. Patients treated with Afatinib and Vinorelbine combination therapy could continue to receive treatment until second progression of disease, intolerable side effects, or withdrawal of consent. The 95% Confidence Interval is Exact Confidence Interval.
Arm/Group | Afatinib Once Daily (OD). Afatinib+V (Vinorelbine).
Number analyzed (Participants) | 26
Days | 253.0 [166.0 to 713.0]

ADVERSE EVENTS:
Time Frame: Part A: From first study drug administration in Part A to last study drug administration in Part A + up to 28 days (max. 728). Part B: From first study drug administration in Part B to last study drug administration in Part B + up to 28 days (max. 265).
Description: The additional 28 days is the residual effect period which was added to the last study drug administration in each part. This may have been truncated in Part A where patients started Vinorelbine prior to the 28 days elapsing.
Groups:
- Part B: Afatinib+V (Vinorelbine).: Part B: Upon first Progression of Disease (PD), patients could enter Part B of the study, during which they continued to be treated with Afatinib and additionally were treated with Vinorelbine 25 mg/m2 per week via intravenous (i.v) infusion. Patients treated with Afatinib and Vinorelbine combination therapy could continue to receive treatment until second progression of disease, intolerable side effects, or withdrawal of consent.
Arm/Group | Part A: Afatinib Once Daily (OD). | Part B: Afatinib+V (Vinorelbine).
Serious Adverse Events (participants affected / at risk) | 12/26 | 4/10
Other Adverse Events (participants affected / at risk) | 26/26 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Afatinib Once Daily (OD). (N=26) | Part B: Afatinib+V (Vinorelbine). (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Afatinib Once Daily (OD). (N=26) | Part B: Afatinib+V (Vinorelbine). (N=10)
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 1 | 8
Atrial flutter (Cardiac disorders) | 0 | 1
Dry eye (Eye disorders) | 3 | 0
Panophthalmitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 23 | 6
Dry mouth (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 7 | 5
Stomatitis (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 7 | 1
Catheter site erythema (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 5
Mucosal inflammation (General disorders) | 10 | 3
Pyrexia (General disorders) | 1 | 2
Abscess limb (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 1
Eye infection (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 9 | 0
Rhinitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 7 | 4
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 10 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 3 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Breast pain (Reproductive system and breast disorders) | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1
Fungating wound (Skin and subcutaneous tissue disorders) | 0 | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 17 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0
Lymphoedema (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Boehringer Ingelheim (BI) decided to stop further inclusion of patients and stop further treatment with the combination of Afatinib and Vinorelbine as of 03-May-2013. Recruitment into the trial was stopped by amendment in Jul 2013.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.